CLINICAL TRIAL: NCT01086904
Title: Etude de Phase II évaluant l'immunogénicité et la tolérance d'un Vaccin inactivé Non adjuvanté Contre la Grippe A (H1N1) après Transplantation rénale
Brief Title: Safety and Efficacy of an Inactivated and Non Adjuvanted Vaccine Against Influenza A in Renal Transplant Recipients
Acronym: Transfluvac
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C09-32; 2009-016659-23 (EudraCT Number)
Record Dates: First submitted 2009-11-16; First posted 2010-03-15 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2010-07

CONDITIONS: Renal Transplant Recipients; Immunosuppression
Keywords: renal transplantation; immunosuppression; inflenza A (H1N1); vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: inactivated non adjuvanted pandemic H1N1 vaccine — two administrations at D and D21 (15 µg HA)

SUMMARY:
The study is aimed at assessing the safety and efficacy of an inactivated and non adjuvanted Influenza A (H1N1) vaccine in renal transplant recipients.

DETAILED DESCRIPTION:
120 renal transplant recipients under triple immunosuppression will be immunized against influenza H1N1v.

The primary endpoint will be the humoral immunity assessed 21 days after each injection on day 0 and day 21:

* seroprotection rate, defined as the percentage of patients with an antibody title against Hemaglutinin ≥ 1/40e after immunization
* seroconversion rate, defined as the the percentage of patients with an antibody title against Hemaglutinin < 1/10e before immunization and ≥ 1/40e after or with a prevaccine title ≥1/10e increasing at least 4 fold after immunization
* seroconversion factor, defined as the ratio between pre and post vaccine geometrical means of the antibody titles.

Secondary endpoints will be:

* Seroconversion rate, seroprotection rate and seroconversion factor on day 182
* Percentage of patients with an antibody title > 1/40e on day 182 (Immune memory)
* Number and severity of clinical and biological adverse events
* Number of cases of pandemic H1N1v influenza virologically confirmed
* Study of associated parameters influencing the results of H1N1v vaccination in terms of seroprotection, seroconversion and seroconversion factor
* Assessment of the cellular immune response against H1N1v
* Assessment of the H1N1v vaccination on graft function and on humoral anti-HLA response.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 and < 60 years old
* Signed information consent
* Social security coverage
* Renal transplantation > 6 months with a creatinine clearance > 20 ml/mn
* Stable renal function defined as serum creatinine variation < 20 % for the last three months
* Receiving a triple immunosuppression regimen including steroids, Calcineurine inhibitors (cyclosporine or Tacrolimus), and IMPDH inhibitors (Mycophenolate Mofetil or mycophenolic acid)
* Regular follow-up

For child bearing aged female:

* Negative urinary HCG
* Contraception during the first three months of the study

Exclusion criteria:

* Poor renal function defined as creatinine clairance < 20 ml/mn
* Unstable renal function defined as serum creatinine variations > 20 % during the last 3 months
* Cellular or humoral acute rejection episode during the last 3 months before inclusion
* Known HIV, HBV or HCV infection
* Other vaccine administered during the last 3 weeks before inclusion or scheduled in the month after the second vaccine injection
* Known allergy to egg proteins or to one the vaccine compounds
* Severe adverse events after prior administration of any influenza vaccine
* Multiple sclerosis
* Past history of Guillain Barre syndrome
* Fever at inclusion
* H1N1 influenza episode with positive virological tests during the last 6 months
* Contact with people infected with H1N1 influenza during the week prior to inclusion
* Cancer requiring radiotherapy or chemotherapy during the last 6 months
* Blood transfusion during the last 3 months
* Pregnancy during the last 3 months
* No follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Specific humoral response 21 days after each administration Seroprotection and seroconversion rates | after each vaccination and at 6 months

SECONDARY OUTCOMES:
Seroprotection and seroconversion rates at day 182;Percentage of patients with anti-H1N1v Antibodies >1/40e at day 182; Number of undesired events and of Influenza A cases; Assessment of cellular immune response against Influenza A H1N1; Effect of vacc | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre hospitalier Lyon Sud, service de néphrologie transplantation, Pierre-Bénite, Lyon
  - Hôpital E. Herriot , Service de néphrologie, transplantation et immunologie clinique, Lyon
  - Service d'urologie, GH Pitié Salpêtrière, Paris